CLINICAL TRIAL: NCT06320717
Title: A Retrospective/Prospective Study of an Artificial Intelligence Derived Histological Biomarker to Select Neoadjuvant Treatment for Patients With Borderline Resectable or Resectable Pancreatic Ductal Adenocarcinoma
Brief Title: AI Derived Biomarker to Select Neoadjuvant Treatment for Borderline Resectable Pancreatic Ductal Adenocarcinoma
Status: Recruiting | Type: Observational
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: I-3574823
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Borderline Resectable (Cohort A): Pathological response of Patients with borderline resectable disease (per NCCD Criteria) treated with standard care chemotherapy
  Interventions: Other: Blood sample
- Patients with Resectable (Cohort B): Pathological response of Patients with resectable disease (per NCCN criteria) treated with standard care chemotherapy
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — To determine if there are any biomarkers in the blood that could be used to choose best treatment plan for future patients

SUMMARY:
To collect samples and information from patients who will be undergoing standard of care neoadjuvant treatment with either FOLFIRINOX or Gemcitabine + Nab-paclitaxel.

The information collected will be used to determine if there are any "biomarkers" in your blood or tumor tissue that, when compared to your response to the neoadjuvant treatment, could be used to choose the best treatment option for future patients with similar biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically confirmed PDAC that is borderline resectable (BR) (Cohort A) OR have histologically or cytologically confirmed PDAC that is resectable (Cohort B) using the National Comprehensive Cancer Network criteria [35].
* Availability of archival tumor tissue (diagnostic for PDAC) required
* Have a documented ECOG Performance Status of ≤ 1
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form (ICF) prior to receiving any study related procedure.

Exclusion Criteria:

* Has received prior systemic treatment (standard of care or experimental) for PDAC
* Participant has a concurrent malignancy requiring active treatment during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community practices and hospital clinics
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2026-07-02 (Estimated); Study Completion 2026-07-02 (Estimated)

PRIMARY OUTCOMES:
Retrospective prediction of pCR in resectable patients | Up to 2 years
  Pathologic response is based on the American College of Pathology Criteria. The AI classified treatment is based on the best representative slide analyzed by the Valar Labs AI algorithm for V-FFX (is Folfirinox recommended) and V-GNP (is GEM/NAB-Paclitaxel recommended
Retrospective prediction of pCR in borderline resectable patients | Up to 2 years
  Pathologic response is based on the American College of Pathology Criteria. The AI classified treatment is based on the best representative slide analyzed by the Valar Labs AI algorithm for V-FFX (is Folfirinox recommended) and V-GNP (is GEM/NAB-Paclitaxel recommended).
  Pathologic response is based on the American College of Pathology Criteria. The AI classified treatment is based on the best representative slide analyzed by the Valar Labs AI algorithm for V-FFX (is Folfirinox recommended) and V-GNP (is GEM/NAB-Paclitaxel recommended)

SECONDARY OUTCOMES:
Survival status | Up to 2 years
  Medical chart will be reviewed for survival status
RECIST 1.1 response | UP to 2 years
  Tumor response was determined by RECIST1.1

CONTACTS AND LOCATIONS:
Overall Officials: Christos Fountilas, MD, Principal Investigator — Roswell Park Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Good Samaritan University Hospital, West Islip, New York